CLINICAL TRIAL: NCT00396604
Title: A Randomized, Double-blind, Double-dummy, Active (Formoterol 12 µg b.i.d) and Placebo Controlled, Multi-center, 5 Period Crossover Study to Assess the Bronchodilatory Efficacy and Safety of Single Doses of Indacaterol 150 µg, 300 µg and 600 µg Delivered Via Single Dose Dry Powder Inhaler vs. Placebo in Patients With Moderate to Severe COPD.
Brief Title: Indacaterol Delivered Via a Single Dose Dry Powder Inhaler (SDDPI) in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149B2212
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; COPD; Lung Diseases, Obstructive
Keywords: indacaterol; long acting beta agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive

INTERVENTIONS:
Drug: indacaterol maleate

SUMMARY:
The study is designed to obtain safety and efficacy data on three dose levels of indacaterol when delivered via an SDDPI in patients with COPD. All patients will receive 1 day of treatment with each of the following: indacaterol 150 µg, once- indacaterol 300 µg, indacaterol 600 µg, placebo, and formoterol. Each treatment day will be followed by a washout-period of 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged 40-75 years with COPD and symptoms such as cough, sputum production, and shortness of breath.
* Smoking history of at least 10 pack years
* FEV1 less than 65% of the predicted normal value and at least 0.75 L
* Pre-bronchodilator FEV1/FVC less than 70%

Exclusion Criteria:

* A history of asthma or COPD diagnosis before the age of 40
* Hospitalization for COPD exacerbation within the previous 6 weeks
* Respiratory tract infection within 6 weeks
* Use of long-term oxygen therapy
* Diabetes type I or uncontrolled diabetes type II
* Clinically relevant laboratory abnormality or clinically significant condition
* Corrected QT interval (QTc) above 430 ms for males and 450 ms for females, or a history of QTc prolongation. Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Lung function measured 24 hours after having taken medication, by a special test called "forced expiratory volume in 1 second "(FEV1)

SECONDARY OUTCOMES:
FEV1 at time points 30 min, 1, 2 and 4hours post-dose
Percent change in FEV1 at time points 30 min, 1, 2 and 4 hours, 23 hours 10min and 23 hours 45 min post dose
Forced vital capacity (FVC) at time points 30 min, 1, 2 and 4 hours, 23 hours 10 min and 23 hours 45 min post dose
Standardized FEV1 area under the curve (AUC) between baseline and 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis
Locations (1):
- Novartis, Vilvoorde, Belgium

REFERENCES:
- [Derived] Hosoe M, Woessner R, Matsushima S, Lawrence D, Kramer B. Efficacy, safety and pharmacokinetics of indacaterol in Caucasian and Japanese patients with chronic obstructive pulmonary disease: a comparison of data from two randomized, placebo-controlled studies. Clin Drug Investig. 2011;31(4):247-55. doi: 10.2165/11586520-000000000-00000. PMID 21184620